CLINICAL TRIAL: NCT06543693
Title: The Development and Assessment of the Core Ultrasound Applications for Nurse Practitioners in Taiwan
Brief Title: The Core Ultrasound Applications for Nurse Practitioners
Status: Active, not recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202112120RINB
Record Dates: First submitted 2024-07-25; First posted 2024-08-09 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Immediate and 3-month Assessment of PoCUS Performance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: ultrasound training — PoCUS training

SUMMARY:
This project aims to establish point-of-care ultrasound (PoCUS) training course for nurse practitioners in Taiwan, and standardized evaluation modules. The study subjects are nurse practitioners across different hospital levels.

I

DETAILED DESCRIPTION:
This project aims to establish point-of-care ultrasound (PoCUS) training course for nurse practitioners in Taiwan, and standardized evaluation modules. The study subjects are nurse practitioners across different hospital levels.

ELIGIBILITY:
Inclusion Criteria:

nursing practitioners who are interested in PoCUS.

Exclusion Criteria:

nursing practitioners who are not interested in PoCUS.

Ages: 20 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: nursing practitioners
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
written test | 1day
  10 multi-choice questionaire
hands-on performance | 1 day
  using 5-point Likert scale. Point 1 indicated no recognizable structures; point 2 indicated minimally recognizable structures but insufficient for diagnosis; point 3 indicated minimal criteria met for diagnosis, recognizable structures but with some technical flaws; point 4 indicated all structures imaged well and diagnosis easily supported; point 5 indicated all structures imaged with excellent image quality and diagnosis completely supported

SECONDARY OUTCOMES:
written test at the 3-month assessment | 3 months
  10 multi-choice questionaire
hands-on performance at the 3-month assessment | 3 months
  using 5-point Likert scale. Point 1 indicated no recognizable structures; point 2 indicated minimally recognizable structures but insufficient for diagnosis; point 3 indicated minimal criteria met for diagnosis, recognizable structures but with some technical flaws; point 4 indicated all structures imaged well and diagnosis easily supported; point 5 indicated all structures imaged with excellent image quality and diagnosis completely supported

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Ching Lien, Principal Investigator — NTUH
Locations (1):
- Wan-Ching Lien, Taipei, Taiwan, Taiwan